CLINICAL TRIAL: NCT02712164
Title: Molecular, Histologic, and Clinical Analysis of Negative Pressure Wound Therapy (NPWT) for Split-thickness Skin Graft (STSG) Donor Sites
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of resources.
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Indranil Sinha, Assistant Professor of Surgery, Harvard Medical School, Division of Plastic Surgery, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016P000030
Record Dates: First submitted 2016-02-29; First posted 2016-03-18 (Estimated); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Split-thickness Skin Graft Donor Sites; Burns
Keywords: Split-thickness skin graft; STSG; donor site; negative-pressure wound therapy; NPWT; dressing
MeSH Terms: conditions — Burns

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Modified NPWT dressing (Experimental): In the experimental group, a microporous silver-impregnated foam with a thin silicone contact layer (Mepilex Ag) will be applied. A macroporous foam layer (V.A.C. GranuFoam) and an occlusive dressing (V.A.C. Drape) will then be applied to cover the foam, plus 3-5cm border of intact skin. The occlusive dressing will then be pinched and a 2cm hole will be cut to apply the SensaT.R.A.C. Pad that supplies pressure from the NPWT unit. NPWT will be applied at 125mmHg throughout treatment using KCI's InfoV.A.C. Therapy Unit. The donor site dressing will be replaced on postoperative day 5-7 and a new occlusive dressing (Tegaderm) will be applied.
  Interventions: Device: Modified NPWT dressing; Device: Tegaderm
- Control: Tegaderm (Active Comparator): In the control group, the donor sites will be dressed with an occlusive dressing only (Tegaderm). The donor site dressings will be replaced on postoperative day 5-7 and a new occlusive dressing (Tegaderm) will be applied.
  Interventions: Device: Tegaderm

INTERVENTIONS:
Device: Modified NPWT dressing — Use of negative pressure wound therapy on split-thickness skin graft (STSG) donor sites
  Arms: Experimental: Modified NPWT dressing
Device: Tegaderm — Standard of care for STSG donor sites.

SUMMARY:
The purpose of this single-center, randomized, prospective cohort study is to evaluate the clinical outcome and negative-pressure wound therapy (NPWT) mediated modulation of the biologic milieu of a modified NPWT dressing on split-thickness skin graft (STSG) donor sites.

DETAILED DESCRIPTION:
The investigators have designed a prospective randomized trial in which subjects will be assigned to a modified negative-pressure wound therapy (NPWT) dressing or standard moist dressing. The investigators will measure the percentage of re-epithelization at set postoperative time intervals using digital photography, pain using the visual analog scale (VAS), and healing quality using the Vancouver Scar Scale (VSS). The investigators hypothesize that the NPWT will lead to less pain and increased re-epithelization in a shorter postoperative time course. This specific aim seeks to prove/disprove that patients who receive a modified NPWT dressing perceive the advantage with improved healing, pain, shorter length of stay, and other wound symptoms related to delayed donor site wound healing.

The donor site for STSGs provides a consistent model of superficial wounds that offers the opportunity to study both mechanisms of wound healing and potential mechanisms of action of NPWT. In patients undergoing both standard dressings and NPWT, the investigators will sample the wound exudate and perform microbiopsies of the healing wound at fixed intervals and perform histologic and molecular analysis in order to quantify the degree of re-epithelization and the trophic and inflammatory profile of the healing wound.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60
* Both genders are eligible for study
* Written consent obtained from the subject or agent
* Donor site wounds must not exceed 5% total body surface area (TBSA)
* Subject must be receiving a split-thickness skin graft (STSG)
* Donor site is amenable to either NPWT or standard of care (occlusive dressing)
* Ability to comply with necessary wound care/follow up

Exclusion Criteria:

* Age <18 years
* Subject has been diagnosed with Diabetes
* Subject is a smoker
* Subject takes steroids
* Subject takes immunosuppressive medications
* Subject with immunosuppressive disorders
* Donor site wounds that exceed 5% total body surface area (TBSA)
* Subject has sensitivity to silver or acrylic adhesives
* Inability to comply with necessary wound care/follow up.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2017-07 (Estimated); Primary Completion 2018-07 (Estimated); Study Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
Pain as measured by visual analog scale (VAS). | Assessed up to 14 days
Wound healing rate (re-epithelialization) | Assessed up to 1 month
  Evaluated by the investigator and by a blinded expert using photographs.
Wound exudate: mRNA expression | Assessed up to 14 days
  Wound exudate and tissue lysate will be subjected to polymerase chain reaction (PCR) for semi-quantitative analysis of mRNA expression.
Wound exudate: protein content | Assessed up to 14 days
  Quantitative enzyme-linked immunosorbent assay (ELISA) will allow analysis of target protein content.
Tissue sample: re-epithelialization and granulation percentage | Assessed up to 14 days
  Tissue samples will be fixed and processed for hematoxylin and eosin (H&E) staining and analyzed microscopically for re-epithelialization percentage.
Tissue sample: epidermal thickness | Assessed up to 14 days
  Tissue samples will be fixed and processed for hematoxylin and eosin (H&E) staining and analyzed microscopically for epidermal thickness.

SECONDARY OUTCOMES:
Wound Healing Quality | Assessed up to 1 month postoperatively
  As measured by the Vancouver scar scale (VAS)

REFERENCES:
- [Background] Genecov DG, Schneider AM, Morykwas MJ, Parker D, White WL, Argenta LC. A controlled subatmospheric pressure dressing increases the rate of skin graft donor site reepithelialization. Ann Plast Surg. 1998 Mar;40(3):219-25. doi: 10.1097/00000637-199803000-00004. PMID 9523602
- [Background] Orgill DP, Bayer LR. Negative pressure wound therapy: past, present and future. Int Wound J. 2013 Dec;10 Suppl 1(Suppl 1):15-9. doi: 10.1111/iwj.12170. PMID 24251839
- [Background] Glass GE, Murphy GF, Esmaeili A, Lai LM, Nanchahal J. Systematic review of molecular mechanism of action of negative-pressure wound therapy. Br J Surg. 2014 Dec;101(13):1627-36. doi: 10.1002/bjs.9636. Epub 2014 Oct 8. PMID 25294112
- [Background] Fischer S, Wall J, Pomahac B, Riviello R, Halvorson EG. Extra-large negative pressure wound therapy dressings for burns - Initial experience with technique, fluid management, and outcomes. Burns. 2016 Mar;42(2):457-65. doi: 10.1016/j.burns.2015.08.034. Epub 2016 Jan 13. PMID 26774601
- [Background] Nuutila K, Siltanen A, Peura M, Harjula A, Nieminen T, Vuola J, Kankuri E, Aarnio P. Gene expression profiling of negative-pressure-treated skin graft donor site wounds. Burns. 2013 Jun;39(4):687-93. doi: 10.1016/j.burns.2012.09.014. Epub 2012 Nov 8. PMID 23141686